CLINICAL TRIAL: NCT04015297
Title: The Role of Raman Spectroscopic Analysis for Endometriosis Diagnosis
Brief Title: Raman Spectroscopy and Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ob&gyn raman
Record Dates: First submitted 2019-07-06; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis; Endometrioma
Keywords: endometriosis; raman analaysis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): healthy controls
  Interventions: Diagnostic Test: raman analysis
- patient (Experimental): patients diagnosed with endometriosis
  Interventions: Diagnostic Test: raman analysis

INTERVENTIONS:
Diagnostic Test: raman analysis — negative or pozitive

SUMMARY:
We aimed to use Raman spectroscopy to detect differences between healthy controls and patients with surgically proven endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease whose molecular basis is still unknown and diagnostic methods are controversial. The diagnosis is still invasive and there are no accepted ways which are molecular-based and noninvasive. Raman spectroscopy is a vibrational spectroscopy technique which can analyze specific spectral patterns, substances and molecular changes with high specificity. We aimed to use Raman spectroscopy to detect differences between healthy controls and patients with surgically proven endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* proven endometriosis

Exclusion Criteria:

* having additional health conditions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females have endometriosis
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic specificity | 2 years
  differentiating endometriosis patients from healthy controls by computer based technology designed with raman data

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Yuksel, md, Study Director — esenler maternity and children's hospital
Locations (1):
- Bahar Yuksel, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
only by request

REFERENCES:
- [Background] Lyng FM, Traynor D, Ramos IR, Bonnier F, Byrne HJ. Raman spectroscopy for screening and diagnosis of cervical cancer. Anal Bioanal Chem. 2015 Nov;407(27):8279-89. doi: 10.1007/s00216-015-8946-1. Epub 2015 Aug 16. PMID 26277185
- [Background] Eberhardt K, Stiebing C, Matthaus C, Schmitt M, Popp J. Advantages and limitations of Raman spectroscopy for molecular diagnostics: an update. Expert Rev Mol Diagn. 2015 Jun;15(6):773-87. doi: 10.1586/14737159.2015.1036744. Epub 2015 Apr 15. PMID 25872466